NCT01911676 Translational Neuroscience Optimization of GlyT1 Inhibitor

**Statistical Analysis Plan** 5/28/2021

## **Statistical Analysis Plan:**

All dependent measures were assessed for normality using normal probability plots. Descriptive statistics were calculated prior to analyses. Each dependent variable was analyzed using a mixed effects model with dose (placebo, low, high), visit (pre- vs. post-drug), their interaction and period (first or second) as main effect. Interactions involving period were also assessed but were dropped from the models for parsimony. Subject was the clustering factor and the best-fitting variance-covariance structure for the repeated measures in each model was selected based on Schwartz' Bayesian Criterion. Least square means and standard errors were calculated to describe the patterns of means for each outcome. Post-hoc mean comparisons were tested to explain significant effects in the models. Additionally, for each outcome effect slices for the interaction are reported although those should be interpreted with caution when there are no significant interactions.